CLINICAL TRIAL: NCT02816294
Title: Housing Prescriptions as Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Project Hope Boston (Unknown); Boston Housing Authority, City of Boston (Unknown); Nuestra Comunidad Community Development Corporation (Unknown); Medical Legal Partnership Boston (Unknown); The Boston Foundation (Unknown); Blue Cross Blue Shield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-35188
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Housing Instability; High Emergency Department Utilization; Medical Complexity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Housing Prescription (Experimental): Participants in the intervention group will be referred to the Care Coordinator at Project Hope, who will conduct case management with the family to stabilize their housing. The Care Coordinator will refer families all families to benefit maximization services and complete Problem Solving Education. The Care Coordinator will also refer families as necessary to Medical-Legal Partnership Boston for pro-bono legal services and/or the Boston Housing Authority for priority on a subsidized housing waitlist.
  Interventions: Behavioral: Housing Prescription
- Resource List (No Intervention): At present, for families facing housing insecurity, Children's HealthWatch offers paper resources with contact information for local social service agencies that may assist with housing stability.

INTERVENTIONS:
Behavioral: Housing Prescription
  Arms: Housing Prescription

SUMMARY:
Housing Prescriptions as Health Care is a research project studying the effects of an innovative intervention that combines services across the health, housing, social and legal service sectors in order to improve housing stability and child health outcomes among participants. The housing intervention developed for this study specifically addresses issues including families who are: paying more than 50 percent of income on rent or utilities, moving frequently, experiencing homelessness, but are not eligible for shelter through the Department of Housing and Community Development's Emergency Assistance program, or were unable to pay rent on time in the past year. This research explores how coordinated and comprehensive housing services offered through intensive case management improves housing stability and health outcomes for families of young children.

DETAILED DESCRIPTION:
Background:

Housing insecurity is a known risk factor for negative child health and developmental outcomes. The goal of this intervention is to reduce housing insecurity among families with young children as a mechanism for improving child health and improving other predictors on the pathway toward child health, including food security and maternal mental health status.

Rationale:

Children's HealthWatch data collected from 2010-2014 at Boston Medical Center, where the sample for this project will be recruited, found 32% of families were behind on rent in the past year and 7% of families moved more than twice in the past year. Previous research by Children's HealthWatch links multiple moves with increased risks of fair or poor child health and developmental delay. Families who are behind on rent are also at risk of fair or poor health, developmental delays, and are below average in length/height, a marker for under-nutrition. Given the significant associations between housing insecurity and child health outcomes, this project is tailored to address challenges faced by families who are severely housing insecure and who are classified as high health care utilizers by industry standards (defined as ≥ 3 emergency department visits in one year).

This research study design for this pilot is a randomized control trial whereby eligible families are randomly assigned to the intervention group or the control group. Those in the intervention group will be referred to a case manager and receive at least one of the six services offered through the program. Families in the control group will receive the current standard of care, which is a packet of outreach resources with information on housing and housing supports.

Purpose:

This study will investigate if this intervention is effective in improving housing stability and child health outcomes compared to current standard of care.

Study hypotheses:

Using data collected at baseline, six months, and 12 months after enrollment, the investigators will examine whether children ages 0-4, their siblings ages 0-11, and caregivers in the intervention group, vs. those in the control group, are more likely to have:

* Reduced score on housing insecurity assessment
* Reduced emergency department (ED) usage and hospitalizations for caregivers and children
* Improved adherence to well-child visits and immunization schedule
* Improved caregiver mental health, as defined by reduced depressive symptoms reported
* Increased family income and reduced reports of material hardships, including decreased food insecurity, defined by the gold-standard USDA 18-item scale; decreased energy insecurity, using the validated Children's HealthWatch screener; and decreased health care hardships, using the Children's HealthWatch screener.

The investigators will also examine ultimate net cost vs. savings per consumer to implement this Housing Prescription as Health Care program. Elements we will consider in economic models include:

* Costs of delivery of the intervention
* Savings from avoided health care costs
* Savings from avoided homelessness
* Increased family income as a result of this intervention

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of family experiencing housing instability
* One or more family members in the household must have had >= 3 emergency room visits in the past year or child with medical complexity enrolled in comprehensive clinical case management program
* Caregiver of child <11 years, who receives primary care at Boston Medical Center

Exclusion Criteria:

* None of the members of the household have had >=3 emergency room visits in the past year nor medically complex child enrolled in case management.
* Family in stable housing
* Index child not a primary care patient at Boston Medical Center
* All children in household >11 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in housing stability | baseline, six months, twelve months, 18 months, 24 months
  Measured using self-report data on frequency of moves, risk of eviction, and rent affordability. Data collected at baseline, six months, and twelve months to assess change in housing stability from baseline at each time point.

SECONDARY OUTCOMES:
Emergency Department utilization | baseline, six months, twelve months, 18 months, 24 months
  Measured using self-report data of number of emergency department visits in the year prior to the study, six months after enrollment, and twelve months after enrollment.
Adherence to well-child visits schedule | one year, two years
  Assessed by successful attendance of well-child visits recommended by the primary care physician and tracked in the electronic health record.
Adherence to immunization schedule | one year, two years
  Assessed by successful completion of vaccinations as recommended by the primary care physician and tracked in the electronic health record.
Caregiver mental health | baseline, six months, twelve months, 18 months, 24 months
  Measured using the Patient Health Questionnaire (PHQ-2) validated screener, which will be administered at baseline, six months, and twelve month.
Food security | baseline, six months, twelve months, 18 months, 24 months
  Measured using the United States Department of Agriculture Food Security Survey Module at baseline, six, and twelve month follow up
Energy security | baseline, six months, twelve months, 18 months, 24 months
  Measured using validated home energy screener from Children's HealthWatch at baseline, six, and twelve months
Health care hardships | baseline, six months, twelve months, 18 months, 24 months
  Measured by self-report of either foregoing health care due to other household expenses or trading off household expenses to pay for health care. Data will be collected at baseline, six, and twelve months.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Sandel, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutts DB, Meyers AF, Black MM, Casey PH, Chilton M, Cook JT, Geppert J, Ettinger de Cuba S, Heeren T, Coleman S, Rose-Jacobs R, Frank DA. US Housing insecurity and the health of very young children. Am J Public Health. 2011 Aug;101(8):1508-14. doi: 10.2105/AJPH.2011.300139. Epub 2011 Jun 16. PMID 21680929
- See also: Children's HealthWatch report on behind on rent — http://www.childrenshealthwatch.org/wp-content/uploads/behindcloseddoors_report_jan11-.pdf